CLINICAL TRIAL: NCT05637619
Title: Natural Dentition, Prosthesis and Antagonist Wear 3D Analysis
Status: Recruiting | Type: Observational
Sponsor: Implantology Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ||2022-11
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Wear, Tooth; Dental Prosthesis Complication; Wear, Occlusal
Keywords: Tooth wear; Full arch Implant; 3D scanner; Prosthesis; Screw retained; Zirconia; Hybrid Acrylic
MeSH Terms: conditions — Tooth Wear; Tooth Attrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dentate Patients: Patients with natural dentition - maxilla and mandible
  Interventions: Behavioral: Dentate Patients
- Zirconia: Patients that have a full-mouth (maxilla or mandible) dental implant supported rehabilitation restored with monolithic zirconia biomaterial
  Interventions: Device: Monolithic Zirconia
- Hybrid Acrylic: Patients that have a full-mouth (maxilla or mandible) dental implant supported rehabilitation restored with acrylic material (hybrid acrylic)
  Interventions: Device: Hybrid-Acrylic

INTERVENTIONS:
Device: Monolithic Zirconia — Maxillary or/and mandibular screw retained zirconia monolithic prostheses supported by at least 4 implants
  Groups: Zirconia
Device: Hybrid-Acrylic — Maxillary or/and mandibular screw retained hybrid prostheses supported by at least 4 implants;
  Groups: Hybrid Acrylic
Behavioral: Dentate Patients — Dentate Patients with natural dentition or tooth supported crowns
  Groups: Dentate Patients

SUMMARY:
Wear resistance is one of the most important physical properties of teeth, and wear resistance of zirconia against artificial acrylic, enamel and composite resin denture teeth has not been clearly established.

Implant-supported dental restorations present a higher threshold for occlusion perception when compared to natural teeth, which can occlusal overload mechanisms or lead to wear of rehabilitation materials or the antagonist arch.

In clinical conditions, however, many other factors influence the complex interaction between dental enamel and opposing substrates: patient-related factors such as dietary habits, dysfunctional occlusion, masticatory forces, and bruxism contribute to accelerated enamel loss of antagonist teeth.

DETAILED DESCRIPTION:
It will be our intention to perform a prospective study and proof-of-concept to assess wear in natural dentition, Full arch implant supported rehabilitation (FAISR) and opposing arches. Wear according to type of rehabilitation and of opposing arch, technical complications, parafunction and number of placed implants will be assessed.

Intra-oral digital acquisition will be performed at pre-defined intervals. Changes over time will be assessed through a previously described digital superimposition methodology volumetric changes determined.

Patients will be scanned using an intraoral dental scanner (T0)

Patients will be recalled at every 4-months (T1), 8-months (T2) and 12-months (T3) visits for re-scanning and from there every 6-months

Scanned images will be compared using a metrology software to determine maximum vertical wear of teeth and root mean square wear.

ELIGIBILITY:
Dentate Group :

Inclusion criteria

* fully dentate (with at least 10 teeth ) and do not have any tooth mobility;
* at least 12months follow up

Exclusion criteria

- missing more than 4 teeth, extensive caries, bonded orthodontic brackets

Edentulous Group:

Inclusion Criteria:

* Maxilla or Mandible Implant full-mouth implant restoration
* Monolithic ceramic or hybrid-acrylic restoration
* at least12 months Follow-up

Exclusion Criteria:

* Heavy bruxists
* Patients that changed the full arch rehabilitation during the study (ex: framework fracture or lab reparation)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Control Group: Healthy Patients, Dentate
  Experimental Groups : Patients from a dental office that did a full-mouth (maxilla or mandible) implant-supported rehabilitation and made the final rehabilitation in either monolithic zirconia or hybrid-acrylic material
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Wear of teeth and materials of restorations | at least 12 months follow-up
  Measure in different groups occlusal tooth wear from insertion (baseline) to 4, 8 and 12 months post-insertion
  Scanned images will be compared using a metrology software to determine maximum vertical wear of teeth and root mean square wear.

SECONDARY OUTCOMES:
Wear of different antagonists | at least 12 months follow-up
  Measure occlusal tooth wear of antagonists from insertion (baseline) to 4, 8 and 12 months post-insertion
  Scanned images will be compared using a metrology software to determine maximum vertical wear of teeth and root mean square wear.

CONTACTS AND LOCATIONS:
Overall Officials: João M Caramês, Phd, Study Director — Implantology Institute; Duarte N Marques, Phd, Study Director — Implantology Institute; Artur F Simões, Msc, Principal Investigator — Implantology Institute
Locations (1):
- Artur Simões, Lisbon, Portugal